CLINICAL TRIAL: NCT03266757
Title: Observational Study of the Clinical Practice in Patients With Borderline Resectable or Resectable or Advanced Pancreatic Adenocarcinoma in Greece
Brief Title: Borderline Resectable or Resectable or Advanced Pancreatic Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Hellenic Society of Medical Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: N/A-NI-PANC-HeSMO-005490
Record Dates: First submitted 2017-07-18; First posted 2017-08-30 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study of the Clinical Practice in patients with Borderline resectable or resectable or advanced pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients Age 18 or older with histologically confirmed ductal pancreatic adenocarcinoma as a primary tumor
* Patients with ductal pancreatic adenocarcinoma (Borderline resectable or resectable or advanced)
* Patients that are alive and under treatment or follow up
* Signed informed consent (ICF)

Exclusion Criteria:

* Presence of other primary tumors
* Pancreatic adenocarcinoma due to metastasis from other primary tumor(s)
* Neuroendocrine or other pancreatic carcinoma other than ductal adenocarcinoma
* Patients who refuse to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Public and Private Hospital Institutions
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2017-02-11 (Actual); Study Completion 2018-02-11 (Actual)

PRIMARY OUTCOMES:
clinical practice-treatments | 2 years

SECONDARY OUTCOMES:
progression Free Survival | 2 years
Overall Survival | 2 years